CLINICAL TRIAL: NCT00680030
Title: Reversibility of Esophageal Dysmotilities Associated With Gastric Banding After Conversion to Gastric Bypass
Brief Title: Reversibility of Dysmotility After Gastric Banding
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: University of Zurich (Other)
Responsible Party: PD Dr. med. Jan Borovicka, MD, Divison of Gastroenterology, Cantonal Hospital St. Gallen
Other Study IDs: EKSG 06/91
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Ineffective Motility; Diffuse Esophageal Spasms; Achalasia-Like Dysmotility
Keywords: impedance; manometry; motility disorders; ineffective motility; diffuse esophageal spasms; achlasia-like dysmotility
MeSH Terms: conditions — Esophageal Spasm, Diffuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
In the current study we plan to evaluate the effects of the conversion from gastric banding to gastric bypass on esophageal function using combined monitoring. The primary aim of the current study is to evaluate esophageal function before and 3-months after the conversion from gastric banding to gastric bypass. A second objective is to evaluate the severity of symptoms, esophageal dysmotilities, endoscopic abnormalities and bolus retention found in patients referred for conversion from gastric banding to gastric bypass. Our hypothesis is that esophageal motility disorders associated with gastric banding are reversed by conversion to gastric bypass.

DETAILED DESCRIPTION:
2.2.3 Research plan

As model for this study we propose a longitudinal single-center study design with testing before and after the surgical intervention.

Participants

The study population will be limited to patients considered for gastric banding to gastric by-pass conversion. Patients will be recruited from the surgical out-patient clinic

Testing during the study period

Pre-OP 3 months post-OP Symptom evaluation X X Endoscopy X X Upper GI series X X Combined MII-EM X X

OP - conversion of gastric band to gastric bypass

After providing informed consent the volunteers will be screened for inclusion/exclusion criteria. Participants fulfilling the inclusion/exclusion criteria will undergo baseline symptom evaluation, endoscopy, an upper GI series and esophageal function testing using combined MII-EM as part of the pre-operative work-up. The same examinations (symptom evaluation, endoscopy, upper GI series and esophageal function testing) will be repeated 3 months after successful conversion from gastric band to bypass.

Symptom evaluation Patients will be asked to complete a standardized esophageal symptom questionnaire. This questionnaire evaluates the frequency and severity of heartburn, chest pain, regurgitation and dysphagia which are then computed into a composite score (Eraflux score ).

Endoscopy Standard sedated endoscopy will be performed by a trained gastroenterologist. The endoscopy will be performed according to the standard clinical protocol. During endoscopy the examiner will pay particular attention to the esophageal mucosa, the size of the gastric pouch above the band (baseline examination), the size of the gastric pouch above the gastro-jejunal anastomosis (post-operative examination), the presence of ulcerations at the site of gastric banding/gastric bypass.

Upper GI Series Patients will undergo upper GI series using a modified timed-barium swallow (achalasia) protocol. Patients will receive 100ml liquid barium and PA images focused on the GE junction will be taken immediately after swallowing, 1 and 3 minutes later. These sequences should allow determining the position of the band relative to the GE junction and the size of the gastric pouch above the gastro-jejunal anastomosis.

Esophageal function testing (EFT)

On the day of esophageal motility testing an EFT probe will be placed transnasally through the esophagus into the stomach and the LES location and pressure will be determined by stationary pull-through technique. The most distal circumferential pressure sensor will be placed in the high-pressure zone (HPZ) of the LES. The other measuring sites (both pressure and impedance) will be subsequently at 5, 10, 15 and 20 cm above the HPZ of the LES. Ten swallows (5 cc each) of liquid (0.9% normal saline) and 10 swallows (5 cc each) of a standard viscous material (EFT viscous, Sandhill Scientific, Inc) will be given with each swallow 20-30 seconds apart.

Analyzed parameters:

* Bolus transit time (BTT): time interval (sec) between bolus entry at the proximal measuring segment and bolus exit at the distal segment
* Smooth muscle bolus transit time (SMBTT): time interval (sec) between bolus entry at the second most distal measuring segment and bolus exit at the distal segment
* Contraction amplitude at 5, 10, 15 and 20 cm above the HPZ
* Distal esophageal amplitude (DEA): average amplitude of contraction at 5 and 10cm above HPZ
* Onset velocity of contractions: contraction velocity between 5 and 10 cm above the HPZ
* LES mid-respiratory resting pressure measured during station pull-through
* Average LES residual pressure during swallowing

Data analysis

Proportions (i.e. percentage of patients with esophageal dysmotility, patients with ulcerations at the banding/anastomosis site, etc.) will be compared using McNemar test. Continuous parameters (i.e. symptom scores, esophageal manometry and bolus transit data) recorded prior and 3-months after the conversion will be compared using paired T-tests. For statistical significance alpha will be set at 0.05.

Sample size calculation Assuming that esophageal dysmotilities are present in 50% of patients prior to the conversion of banding to bypass and that conversion reduces this proportion by 50% we calculated that 40 complete datasets would be required for an 85% power to identify this change. Allowing a drop-out rate of 20% we plan to enroll 50 patients in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom a conversion from gastric band to gastric bypass is planed

Exclusion Criteria:

* Acute cardiac or pulmonary conditions
* Antireflux surgery or antireflux endoscopic procedures.
* Patients unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients in whom a conversion from gastric band to gastric bypass is planed
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-09 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
reversibility of dysmotility after surgery | 3 months

SECONDARY OUTCOMES:
degree of dysmoztility after gastric banding | not defined

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Kuenzler, study nurse, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

REFERENCES:
- [Derived] Borovicka J, Krieger-Grubel C, van der Weg B, Thurnheer M, Schultes B, Sulz MC, Gutzwiler JP, Bisang P, Pohl D, Fried M, Meyenberger C, Tutuian R. Effect of morbid obesity, gastric banding and gastric bypass on esophageal symptoms, mucosa and function. Surg Endosc. 2017 Feb;31(2):552-560. doi: 10.1007/s00464-016-4996-5. Epub 2016 Jun 10. PMID 27287911